CLINICAL TRIAL: NCT04570332
Title: Phase 2 Single Arm Clinical Study to Evaluate the Efficacy and Safety of Intratumoral Administration of BO-112 in Combination With Pembrolizumab in Subjects That Have Progressed on Anti-PD-1-based Therapy for Stage III or IV Melanoma
Brief Title: BO-112 With Pembrolizumab in Unresectable Malignant Melanoma
Acronym: SPOTLIGHT203
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Highlight Therapeutics (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BOT112-03; 2020-003921-51 (EudraCT Number); KEYNOTE-B77 / MK-3475-B77 (Other Grant/Funding Number: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2020-09-22; First posted 2020-09-30 (Actual); Results first posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Melanoma
Keywords: BO112; Intratumoral; Immunotherapy; TLR3; Melanoma
MeSH Terms: conditions — Melanoma | interventions — BO-112; pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is a phase 2 study with one single treatment arm (BO-112 in combination with pembrolizumab)
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Patients will be treated with a combination of IT BO-112 and IV pembrolizumab.BO-112 will be administered once weekly (QW) for the first 7 weeks and then once every three weeks (Q3W); pembrolizumab Q3W will be administered IV. BO-112 will be administered IT at a total dose of 1-2 mg at each administration to 1-8 tumor lesions.
  Interventions: Drug: BO-112 plus pembrolizumab; Procedure: Tissue Biopsies

INTERVENTIONS:
Drug: BO-112 plus pembrolizumab — Patients will be treated with the combination of BO-112 and pembrolizumab. Order of administration should be pembrolizumab then IT BO-112. BO-112 will be administered IT at a total dose of 1-2 mg at each administration to 1-8 tumor lesions using tuberculin (TB) syringes (or equivalent) with 20- to 25-gauge needles
  Other Names: KEYTRUDA®
Procedure: Tissue Biopsies — Pre and post (if feasible) treatment tumor tissue biopsies will be used for correlative research.

SUMMARY:
This is a phase 2, single arm, open label, adaptive design study to determine the preliminary anti-tumor activity and confirm the safety of IT BO-112 in combination with intravenous (IV) pembrolizumab. The study will enroll patients with advanced and/or metastatic melanoma that have progressed on anti-PD-1-containing treatment.

DETAILED DESCRIPTION:
Patients with advanced Stage III/IV melanoma, refractory or resistant to anti-PD-1 treatment, were treated with the combination of intra-tumoral (IT) BO-112 and Q3W IV pembrolizumab. IT administration of BO-112 was performed once weekly (QW) for the first 7 weeks and then once every three weeks (Q3W).

The primary and secondary endpoints include overall response rate (ORR), durability of response (DOR), disease control rate (DCR), progression free survival (PFS), overall survival (OS), and safety profile.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to give written informed consent for the study.
2. Be ≥ 18 years of age on day of informed consent.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Histologically or cytologically confirmed diagnosis of cutaneous or mucosal melanoma.
5. Known BRAF status.
6. Have unresectable stage III or stage IV melanoma. Patients must have progressed on treatment with an anti-PD-1/L1 monoclonal antibody (mAb) administered as monotherapy, or in combination with other checkpoint inhibitors or other therapies. PD-1 treatment progression is defined by meeting all of the following criteria:

   1. Received at least 6 weeks of standard dosing of an approved anti-PD-1/L1 mAb.
   2. Demonstrated disease progression (PD) on or after PD-1/L1 as defined by RECIST v1.1. The initial evidence of PD is to be confirmed by a second assessment no less than four weeks from the date of the first documented PD, in the absence of rapid clinical progression.
   3. Progressive disease documented within 12 weeks from the last dose of anti-PD-1/L1 mAb.

   i. This determination is made by the investigator. Once PD is confirmed, the initial date of PD documentation will be considered the date of disease progression.
7. Anti-PD-1-based therapy should have been the last line of systemic therapy as part of first line treatment. Prior treatment either in neo or adjuvant setting is allowed (if patient did not develop progressive disease while on receiving it). In the case of patients who develop progressive disease during adjuvant therapy, that treatment will be counted as one prior line, and will be eligible if only that prior line has been administered.
8. At least one tumoral lesion that is RECIST 1.1 measurable and amenable for IT injection.
9. At least one accessible tumor lesion that is amenable to weekly injection. If liver is a site of injection, presence of at least one additional tumor lesion outside the liver amenable for injection.
10. Willingness to provide biological samples required for the duration of the study including a fresh tumor biopsy sample. NOTE: If possible, the biopsied lesion should be a non-target lesion.
11. Adequate hematologic and organ function defined by the following laboratory results obtained within 2 weeks prior to the first dose of study treatment:

    1. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
    2. Platelet count ≥ 100 x 10^9/L
    3. Hemoglobin (Hgb) ≥ 9 g/dL
    4. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5x upper limit of normal (ULN) (5 × ULN if presence of liver metastases)
    5. Serum total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN
    6. Prothrombin time (PT) (or international normalized ratio [INR]) within normal limits and activated partial prothrombin time (aPTT) within normal limits
    7. Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 30 mL/min (calculated per institutional standard)
12. Female patient of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the injection of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
13. Female patients who are not pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment.

    Female patients of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity from the beginning of the study through 120 days after receiving the last dose of study medication. Patients of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.

    Non-pregnant, non-breast-feeding women may be enrolled if they are willing to use 2 methods of birth control or are considered highly unlikely to conceive. Highly unlikely to conceive is defined as 1) surgically sterilized, or 2) postmenopausal (a woman who is ≥45 years of age and has not had menses for greater than 1 year will be considered postmenopausal), or 3) not heterosexually active for the duration of the study. The two birth control methods can be either: two barrier methods or a barrier method plus a hormonal method to prevent pregnancy.
14. Patients should be informed that taking the study medication may involve unknown risks to the fetus (unborn baby) if pregnancy were to occur during the study. In order to participate in the study, they must adhere to the contraception requirement (described above). If there is any question that a patient will not reliably comply with the requirements for contraception, that patient should not be entered into the study.
15. Male patients should agree to use an adequate method of contraception from the beginning of the study through 120 days after receiving the study medication.
16. In countries where human immunodeficiency virus (HIV) positive patients can be included, HIV infected participants must be on anti-retroviral therapy (ART) and have a well-controlled HIV infection/disease defined as:

    1. Participants on ART must have a CD4+ T-cell count >350 cells/mm3 at time of screening;
    2. Participants on ART must have achieved and maintained virologic suppression defined as confirmed HIV RNA level below 50 copies/mL or the lower limit of qualification (below the limit of detection) using the locally available assay at the time of screening and for at least 12 weeks prior to screening;
    3. Participants on ART must have been on a stable regimen, without changes in drugs or dose modification, for at least 4 weeks prior to study entry (Day 1).
17. Able and willing to comply with study and follow-up procedures.

Exclusion Criteria

1. Uveal melanoma.
2. Prior grade 3-4 irAE due to immune checkpoint inhibitors requiring systemic steroids for more than 2 weeks.
3. Prior intra-tumoral treatments.
4. If a liver lesion is the site of injection:

   1. macroscopic tumor infiltration by the lesion to be injected into the main portal vein, hepatic vein or vena cava;
   2. portal vein thrombosis;
   3. prior embolization of liver lesions;
   4. radiofrequency, cryotherapy or microwave ablation in the last 6 months;
   5. Child-Pugh B or C;
   6. All AST, ALT and bilirubin greater than >2.5 ULN.
5. Contraindications to tumor biopsy and injections of the metastasis(es), such as coagulopathy, therapeutic dose anticoagulant treatment and treatment with long-acting agents such as clopidogrel which cannot be safely stopped.
6. Chemotherapy or biological cancer therapy within 4 weeks prior to the first dose of study treatment. Note: Participants must have recovered from all adverse events (AEs) due to previous therapies to ≤ Grade 1 or baseline. Participants with ≤ Grade 2 neuropathy may be eligible.
7. Palliative radiotherapy within 1 week of start of study treatment. Subjects must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
8. Clinically active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
9. History of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years.
10. Allergy to BO-112 and/or any of its excipients.
11. Allergy to pembrolizumab and/or any of its excipients.
12. Active infection requiring systemic therapy.
13. History of (non-infectious) pneumonitis/interstitial lung disease that required steroids or current pneumonitis/interstitial lung disease.
14. Active autoimmune disease that required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
15. Receiving systemic immunosuppressive therapy within 28 days before enrolment with the exceptions of intranasal, topical, and inhaled corticosteroids or oral corticosteroids at physiological doses not exceeding 10 mg/day of prednisone or equivalent.
16. HIV-infected participants with a history of Kaposi sarcoma and/or Multicentric Castleman Disease.
17. Known history of hepatitis B (defined as HbsAg reactive) or known active hepatitis C (defined as HCV RNA [qualitative] detected) virus infection. Patients who are hepatitis B surface antigen negative and HBV viral DNA negative are eligible.

    1. Patients who had HBV but have received an antiviral treatment and show non-detectable viral DNA for 6 months are eligible.
    2. Patients who are seropositive because of HBV vaccine are eligible.
    3. Patients who had HCV but have received an antiviral treatment and show no detectable HCV viral DNA for 6 months are eligible.
18. Has received a live vaccine within 28 days prior to the first dose of study drug. For COVID vaccines a 72 hour wash out period is necessary.
19. History of allogenic tissue or solid organ transplant.
20. Is currently participating or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment (patients who are in a follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent).
21. Any clinically significant psychiatric, social, or medical condition that, in the opinion of the Investigator, could increase patient's risk, interfere with protocol adherence, or affect a patient's ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2024-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marisol Quintero, PhD, Study Director — Highlight Therapeutics
Locations (19):
- France (7):
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Centre Hospitalier Universitaire de Grenoble, Grenoble
  - Hopital Lyon Sud, Lyon
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Centre Hospitalier Universitaire de Nice, Nice
  - Hôpital Ambroise-Paré, Paris
  - Institut Gustave Roussy, Paris
- Spain (12):
  - H. Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - H. Universitari Quirón Dexeus, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Clara Campal - HM Sanchinarro, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Clínica Universidad de Navarra, Pamplona
  - Hospital Universitario Virgen Macarena, Seville
  - H. General Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marquez-Rodas I, Dutriaux C, Saiag P, de la Cruz Merino L, Castanon Alvarez E, Robert C, Rodriguez-Moreno JF, Arance A, Cerezuela-Fuentes P, Montaudie H, Sanmamed MF, Gonzalez-Cao M, Charles J, Lopez Criado MP, Berrocal A, de Miguel E, Funck-Brentano E, Prey S, Alamo de la Gala MC, Melero I, Aviles-Izquierdo JA, Roman R, Garcia-Pelaez B, Rodriguez S, Trnkova ZJ, Quintero M, Macia S, Chaney MF, Dalle S. BO-112 Plus Pembrolizumab for Patients With Anti-PD-1-Resistant Advanced Melanoma: Phase II Clinical Trial SPOTLIGHT-203. J Clin Oncol. 2025 Sep;43(25):2806-2815. doi: 10.1200/JCO-24-02595. Epub 2025 Jun 27. PMID 40577656

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: Patients with advanced Stage III/IV melanoma, refractory or resistant to anti-PD-1 treatment, were treated with the combination of intra-tumoral (IT) BO-112 and Q3W IV pembrolizumab. IT administration of BO-112 was performed once weekly (QW) for the first 7 weeks and then once every three weeks (Q3W).
Period: Overall Study
Arm/Group | Single Arm
Started | 42
Completed | 42
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: Patients with advanced Stage III/IV melanoma resistant or refractory to anti-PD-1 treatment were treated with the combination of IT BO-112 and pembrolizumab. IT administration of BO-112 was performed once weekly (QW) for the first 7 weeks and then once every three weeks (Q3W); pembrolizumab Q3W was administered IV.
Arm/Group | Single Arm
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.67 (15.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  France | 17
  Spain | 25

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Percentage of patients achieving a complete response (CR) or partial response (PR) as best overall response, by independent radiological central review (IRCR) per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: From the first dose of study treatment to the date of CR or PR assessed up to 2 years
Population: Modified intent-to-treat population - patients with baseline and at least one post-baseline assessment. 2 patients from the ITT did not have post-baseline assessment and were excluded from mITT.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Single Arm: Patients were treated with the combination of IT BO-112 and pembrolizumab. IT administration of BO-112 was performed once weekly (QW) for the first 7 weeks and then once every three weeks (Q3W); pembrolizumab Q3W was administered IV.
Arm/Group | Single Arm
Number analyzed (Participants) | 40
percentage of participants | 25.0 [12.69 to 41.20]
Statistical Analysis 1: Comparison: Single Arm; The null hypothesis was H0: ORR=10% (p0) and was tested against H1: ORR>10% at one-sided 5% significance level. Assuming an effect size of ORR=25% (pA), 40 participants provided a power of at least 80%. The minimal statistically significant ORR was 20%; Test type: Superiority; p < 0.01, one-sided test for binomial endpoint; rate % = 25, 95% CI 2-sided [12.69 to 41.20]

2. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: The National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), v5.0 was used for grading toxicities.
Time Frame: 2 years and 9 months
Measure: Count of Participants; unit: Participants
Groups:
- Single Arm: Patients were treated with combination of IT BO-112 and pembrolizumab. IT administration of BO-112 was performed once weekly (QW) for the first 7 weeks and then once every three weeks (Q3W); pembrolizumab Q3W was administered IV.
Arm/Group | Single Arm
Number analyzed (Participants) | 42
Participants | 42

3. Secondary Outcome: Disease Control Rate
Description: Participants with complete response (CR), or partial response (PR), or stable disease (SD) per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR) and modified RECIST 1.1 for immune-based therapeutics (iRECIST)
Time Frame: From the first dose of study treatment to the date of best response (i.e. CR, PR, or SD) on study up to 2 years
Population: 2 participants did not have post-baseline imagining and were excluded from the mITT analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Arm
Number analyzed (Participants) | 40
percentage of participants | 67.5 [50.87 to 81.43]

4. Secondary Outcome: Duration of Response
Description: Median DOR (CR or PR) per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR) by IRCR
Time Frame: From the date of CR or PR until the date of event or censoring up to 2 years
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Single Arm: Patients with advanced Stage III/IV melanoma refractory or resistant to anti-PD-1 treatment were treated with the combination of intra-tumoral (IT) BO-112 and pembrolizumab. IT administration of BO-112 was performed once weekly (QW) for the first 7 weeks and then once every three weeks (Q3W); pembrolizumab Q3W was administered IV.
Arm/Group | Single Arm
Number analyzed (Participants) | 42
months | NA [8.31 to NA] — Median DOR could not be determined by the end of the study due to insufficient number of participants with events

5. Secondary Outcome: Progression Free Survival
Description: Progressive disease (PD) per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR) by IRCR or death
Time Frame: From the first dose of study treatment to the date of radiologic progression or death, whichever comes first, up to 2 years
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Single Arm
Number analyzed (Participants) | 42
months | 3.71 [2.17 to 9.23]

6. Secondary Outcome: Overall Survival
Description: Median overall survival for all patients treated with at least one dose of the study drug
Time Frame: From the first dose of study treatment to death from any cause up to 2 years
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Single Arm: Patients be treated with a combination of IT BO-112 and IV pembrolizumab.BO-112 will be administered once weekly (QW) for the first 7 weeks and then once every three weeks (Q3W); pembrolizumab Q3W will be administered IV. BO-112 will be administered IT at a total dose of 1-2 mg at each administration to 1-8 tumor lesions.
Arm/Group | Single Arm
Number analyzed (Participants) | 42
months | NA [9.89 to NA] — Median could not be determined at the time of study end due to insufficient number of participants with events

ADVERSE EVENTS:
Time Frame: 2 years and 9 months
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 7/42
Serious Adverse Events (participants affected / at risk) | 15/42
Other Adverse Events (participants affected / at risk) | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=42)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) — required hospitalization
Device related infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Condition aggravated (General disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Cerebral hematoma (Nervous system disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Tracheal compression (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=42)
Asthenia (General disorders) | 29 (75)
Pyrexia (General disorders) | 19 (90)
Diarrhoea (Gastrointestinal disorders) | 18 (30)
Nausea (Gastrointestinal disorders) | 13 (32)
Vomiting (Gastrointestinal disorders) | 13 (27)
Chills (General disorders) | 12 (25)
Headache (Nervous system disorders) | 11 (17)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (14)
Decreased apetite (Gastrointestinal disorders) | 10 (13)
Injection site pain (General disorders) | 10 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (14)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (17)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (13)
Oedema peripheral (General disorders) | 7 (9)
Rash (Skin and subcutaneous tissue disorders) | 7 (11)
Constipation (Gastrointestinal disorders) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Hypertension (Vascular disorders) | 6 (8)
Insomnia (Psychiatric disorders) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (9)
Aspartate aminotransferase increased (Investigations) | 5 (6)
COVID-19 (Infections and infestations) | 5 (7)
Influenza like illness (Infections and infestations) | 5 (12)
Dry mouth (Gastrointestinal disorders) | 4 (4)
General physical health deterioratio (General disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Adrenal insufficiency (Endocrine disorders) | 3 (5)
Alanine aminotransferase increased (Investigations) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 3 (4)
Blood alkaline phosphatase increased (Investigations) | 3 (6)
Eye pruritus (Eye disorders) | 3 (3)
Fatigue (Gastrointestinal disorders) | 3 (5)
Gamma-glutamyltransferase increased (Investigations) | 3 (4)
Stomatitis (Gastrointestinal disorders) | 3 (4)
Tremor (Nervous system disorders) | 3 (5)
Vision blurred (Eye disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT04570332/Prot_SAP_000.pdf